CLINICAL TRIAL: NCT03514251
Title: Study on Application of Suturing Parathyroid Markers in Thyroid Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bo Wang,MD (Other)
Responsible Party: Sponsor-Investigator, Bo Wang,MD, Clinical Professor, Fujian Medical University
Organization: Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PT Marker
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Thyroid Cancer; Hypoparathyroidism; Marker; Structural; Complication of Surgical Procedure; Parathyroid Function Low Adverse Event
Keywords: Thyroid Cancer; Hypoparathyroidism; parathyroid marker
MeSH Terms: conditions — Thyroid Neoplasms; Hypoparathyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Routine thyroidectomy and central lymph node dissection
- Parathyroid marker group (Experimental): When the lower parathyroid gland is first seen, the parathyroid gland is sutured with a suture during the operation, and then during this subsequent cleaning, rapid parathyroid localization and parathyroid glands are performed through this marker.
  Interventions: Procedure: The suture marks the location of the parathyroid gland

INTERVENTIONS:
Procedure: The suture marks the location of the parathyroid gland — When the lower parathyroid gland is first seen, the parathyroid gland is sutured with a suture during the operation, and then during this subsequent cleaning, rapid parathyroid localization and parathyroid glands are performed through this marker. Vascular protection.
  Arms: Parathyroid marker group

SUMMARY:
To study the protective effect of suture parathyroid marker method on the function of parathyroid gland in thyroid cancer surgery

DETAILED DESCRIPTION:
This is a prospective randomized controlled study.In the experimental group, the suture parathyroid marker method was used to mark the parathyroid gland at the first time when it shows, and this marker was further used to identify and locating the inferior parathyroid marker in subsequent central region dissection. In the control group, the central area was routinely cleaned without suture parathyroid marker .

ELIGIBILITY:
Inclusion Criteria:

* Patients with thyroid cancer who need central compartment dissection
* Routine neck incision surgery
* Patients undergoing primary neck surgery

Exclusion Criteria:

* Benign thyroid tumor patients
* Selecting patients with endoscopes, small incisions, or robotic surgery
* Patients with hyperparathyroidism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
The stitch marking operation time | During surgery
  The time required for making a parathyroid marker by a suture method
Specimen inspection time | During surgery
  The time required for finding parathyroid glands in surgical specimens
The number of transplanted parathyroid glands | When the surgery is completed
  The number of parathyroid glands required for autotransplantation of parathyroid glands
Parathyroid hormone level testing | 0 days, 1 day, 2 weeks after surgery
  Parathyroid hormone levels before and after surgery
Calcium levels | 0 days, 1 day, 2 weeks after surgery
  Calcium level before and after surgery to detect

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No